CLINICAL TRIAL: NCT00596674
Title: Health Promotion for Women With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2002-08-0043; R01HD035047 (NIH)
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Fibromyalgia
Keywords: Women; Fibromyalgia Syndrome; Health Behaviors; Quality of Life
MeSH Terms: conditions — Fibromyalgia; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle Counts Intervention (Experimental): A wellness intervention that includes 8 weeks of behavior change classes focused on acquiring the skills and knowledge to improve health behaviors (e.g., exercise, stress management), followed by 3 months of phone support.
  Interventions: Behavioral: Lifestyle Counts
- Attention Countrol (Placebo Comparator): 8 weeks of general health classes followed by phone calls for 3 months
  Interventions: Other: Attention Control

INTERVENTIONS:
Behavioral: Lifestyle Counts — 8 weeks of classes focused on health behavior change, individualized goal setting and 3 months of follow-up phone support
  Arms: Lifestyle Counts Intervention
Other: Attention Control — 8 weeks of classes on general health information topics followed by 3 months of phone calls to solicit questions
  Arms: Attention Countrol

SUMMARY:
Women with chronic disabling conditions such as fibromyalgia syndrome (FMS) must manage a wide variety of disease-related, intrapersonal, and environmental demands to maintain their health and quality of life. Engaging in health-promoting behaviors is one strategy recommended to manage disease symptoms and enhance quality of life (USDHHS, 2000). The purpose of this four-year study is to refine and test a theoretically and empirically based intervention to promote the health and well being of women with the chronic disabling condition of fibromyalgia. We hypothesize that women who participate in the "Lifestyle Counts" Intervention will report more greater self-efficacy for health behaviors, more frequent health behaviors and more positive health and quality of life than women in the comparison group.

DETAILED DESCRIPTION:
This wellness intervention, originally developed and tested in a randomized clinical trial of women with MS (N=113), resulted in significant improvements in self-efficacy, health behaviors and improvements in pain, social functioning, mental health and emotional role-functioning. The specific aims of this study are to examine the effects of the adapted wellness intervention on self-efficacy, resources, barriers, health behaviors and health outcomes for women with fibromyalgia.

A sample of 160 women with FMS will be recruited to participate in a randomized clinical study to determine the effects of this wellness intervention that includes an eight week health promotion/behavior change component and 3 months of follow-up phone support. Content regarding stress management, lifestyle adjustment, physical activity, nutrition and women's health issues will be presented with an emphasis on the unique adaptations and associated skills required to empower women with the tools for exercising personal control over their health behaviors. The effects of the intervention on outcome variables will be assessed over an 8-month period with measurements at baseline, 2 months (immediately after the educational/skill-building component), 5 months (after 3 months of phone support) and at 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Physician verified diagnosis of Fibromyalgia for at least 6 months, age 18 to 75,
* Able to speak and read English
* Willing to participate in 8-month intervention study

Exclusion Criteria:

* Pregnancy
* Male
* Concurrent medical conditions (as judged by their physician) for which changes in diet and exercise would be contraindicated

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2003-07; Primary Completion 2007-01 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
SF36 Subscales | Baseline, 2 months, 5 months and 8 months

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire | Baseline, 2 months, 5 months, 8 months
Health Behaviors - The Health Promoting Lifestyle Questionnaire | Baseline, 2 months, 5 months 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexa Stuifbergen, PhD, RN, Principal Investigator — The University of Texas at Austin School of Nursing
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States